CLINICAL TRIAL: NCT04788277
Title: Investigation Into Detection of Prostate Cancer Using Voided Urine
Brief Title: Detection of Prostate Cancer Using Voided Urine
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20G.196; JT 15161 (Other: JeffTrial Number)
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (biospecimen collection): Patients undergo collection of urine samples at baseline during standard of care office/clinic visit.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This study collects urine from male patients seen at the urology clinic to detect prostate cancer cells, shed in voided urine, using the optical imaging method developed in the laboratory, which targets certain biomarkers expressed on prostate cancer cells. The information learned from this study may allow researchers develop a simple diagnostic test for the management of those patients who have elevated prostate specific antigen (PSA) and are suspected to have prostate cancer. It may also help researchers understand the genetic risk factors associated with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To detect prostate cancer cells, shed in voided urine, using the optical imaging method developed in our laboratory, which targets vasoactive intestinal polypeptide receptor 1 (VPAC1) receptors expressed on prostate cancer cells and validates the results with prevailing condition of the patients/volunteers and evaluate diagnostic accuracy.

SECONDARY OBJECTIVES:

I. To establish if the malignant cells as a percent of total cell shed in the urine.

II. To establish the fluorescence intensity around malignant cells. III. To establish if the VPAC protein quantity in shed malignant cells correlate with the aggressiveness of the disease.

OUTLINE:

Patients undergo collection of urine samples at baseline during standard of care office/clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Male
* Patients must be 50-70 years of age
* Willing to comply with all study procedures
* Prior to digital rectal exam (DRE)
* Patients with the diagnosis of prostate cancer (Cohort 1 N=150)

  * Prior to radical prostatectomy/radiotherapy (XRT) or systemic therapy
  * May be on active surveillance
* Patients with elevated PSA level but no know prostate cancer (Cohort 2 N=150)

  * Diagnosis of BPH/lower urinary tract symptoms (LUTS)
  * No prior diagnosis of prostate cancer
  * Prior negative biopsy with PSA > 1.5
  * Without biopsy PSA < 1.5
* Patients with normal PSA levels (Cohort 3 N=200)

  * No documented history of BPH (no medical management or prior surgical treatment for BPH)
  * PSA < 1.5
  * No documented history of prostate cancer
  * No documented history of urothelial carcinoma
* Patients Pre DRE and Post DRE (Cohort 4 N=200)**
* Patients on with a known Gleason Score (Cohort 5= 150)

Exclusion Criteria:

• Patients under the age of 50

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients diagnosed with prostate cancer, male patients with elevated PSA level but no known prostate cancer, and male patients with normal PSA levels and no known prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the vasoactive intestinal polypeptide receptor (VPAC) assay diagnosis | Up to 2 years
  The diagnostic properties of the assay will be assessed by estimating the sensitivity, specificity and positive and negative predictive values, along with their exact Clopper-Pearson 95% compatibility intervals. Subgroup estimates of specificity, positive and negative predictive values and exact compatibility intervals will be generated for comparisons between controls with and without benign prostatic hyperplasia (BPH). All study variables will be summarized and tabulated by prostate cancer status, BPH status, and by percent malignant cells (%M), fluorescence intensity, and VPAC protein quantity. Continuous variables will be summarized in groups by means with standard deviations or, of skewed, by medians with first and third quartiles and with other continuous variables by correlation coefficients. Discrete variables will be summarized by frequency counts and percentages.

SECONDARY OUTCOMES:
Correlations and expected values of aggressiveness | Up to 2 years
  Spearman's correlation coefficients of aggressiveness (measured by Gleason score or prognostic grade group [PGG]) associated with increasing levels of %M, fluorescence intensity, and VPAC protein quantity will be estimated along with 95% compatibility intervals. Linear regression modeling will be used to evaluate how expected values of aggressiveness (measured by Gleason score or PGG are associated with increasing levels of %M, fluorescence intensity, and VPAC protein quantity, respectively, while adjusting for demographics or other study variables that appear to be confounders in preliminary summary analyses. Analyses will be conducted using SAS version 9.4.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Thakur, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No